CLINICAL TRIAL: NCT01317121
Title: Multi-site Communication Deficits Underlying Cognitive Dysfunction in the Prodromal Phase and First Episode of Schizophrenia
Brief Title: Multi-site Communication Deficits in Schizophrenia
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, CMulert, PI, Universitätsklinikum Hamburg-Eppendorf
Other Study IDs: NeuroSFB-PV3632
Record Dates: First submitted 2011-03-15; First posted 2011-03-17 (Estimated); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Schizophrenia; Psychosis
Keywords: Patients with a first episode of schizophrenia; Subjects at risk for psychosis
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Subjects at risk for psychosis: Identification and clinical characterization of subjects with prodromal symptoms will be done in the early diagnosis outpatient center of the University Department of Psychiatry in Hamburg, Germany. Subjects At Risk Mental State (ARMS) for psychosis will be identified if they meet the criteria of the Structured Interview for Prodromal Syndromes (SIPS) (McGlashan et al 2001).
- Patients with a first episode of schizophrenia: Patients with a first episode of schizophrenia will be recruited from inpatients at the Clinic for Psychiatry and Psychotherapy at the University Hospital (UKE) in Hamburg, Germany. All patients have to meet criteria for DSM-IV and ICD-10 diagnosis for schizophrenia.
- Healthy control subjects: Healthy control subjects will be recruited from the hospital staff and students at the University Hospital Hamburg-Eppendorf (UKE), Hamburg, Germany. They have to be free from any neurological or psychiatric disorder, according to DSM-IV and ICD-10 criteria.

SUMMARY:
Multi-site Communication Deficits Underlying Cognitive Dysfunction in the Prodromal Phase and First Episode of Schizophrenia

DETAILED DESCRIPTION:
Abnormal long-range connectivity between brain areas and corresponding impaired synchronization of oscillatory rhythms in neuronal networks represent an important pathophysiological mechanism underlying schizophrenia. Although schizophrenia is considered as a neurodevelopmental disorder the mechanisms by which the abnormal neural circuitry and communication develops before the onset of clinical symptoms are unknown. This project aims to investigate the relationship between disturbed neural synchronization and cognitive deficits in the prodromal phase of schizophrenia and is intended to identify patients with increased risk for developing schizophrenia. Present approaches to describe subjects at risk for psychosis based on clinical features have not been completely convincing since psychiatric symptoms in the prodromal phase are often too unspecific. Recent studies suggest that detecting cognitive deficits might help for a more precise identification of high risk subjects. However, the underlying neurophysiological mechanisms have not yet been investigated sufficiently. Precise identification of subjects with high risk for switching to schizophrenia would be very important since interventional strategies such as medical treatment even with second generation antipsychotics are not completely free of risk and therefore should be limited to subjects with a maximal benefit. In this project subjects at risk for psychosis will be investigated with electroencephalography (EEG), magnetoencephalography (MEG) and simultaneous electroencephalography-functional magnetic resonance imaging (EEG-fMRI). Follow up investigations will be performed after switching to schizophrenia has occurred or not. Neural synchronization between the prefrontal cortex and the hippocampal formation will be investigated using a working memory paradigm. Here, different levels of memory load will be investigated using the n-back paradigm. Earlier studies showed disturbed functional and effective connectivity between the hippocampus and the prefrontal cortex both in patients with schizophrenia and subjects at risk. Neural synchronization between the prefrontal cortex and sensory areas will be investigated with different attentional paradigms. Here, tones will be presented that have to be responded to by button press. Earlier studies demonstrated disturbed auditory evoked gamma oscillations in patients with schizophrenia and unaffected siblings. Neural oscillations will be recorded with 64-channel EEG and localized by means of simultaneous functional magnetic resonance imaging (fMRI). Integration of EEG and fMRI will be performed using single-trial coupling in order to detect brain regions involved in specific oscillatory rhythms. Using both paradigms, neural long-range synchronization will be analyzed. In addition, dynamic causal modelling will be used for further characterization of functional relationships among brain regions involved. The investigators expect a functional relationship between cognitive deficits in subjects with prodromal schizophrenia and subjects with a first episode of schizophrenia with regards to long range neural synchronization. In addition, the investigators expect to identify subjects at high risk for schizophrenia with the analysis of disturbed long range synchronization.

ELIGIBILITY:
Inclusion criteria schizophrenic patients:

* Signed written informed consent.
* Inpatients of the Clinic for Psychiatry and Psychotherapy of the University Hospital Hamburg-Eppendorf (UKE), Hamburg, Germany.
* Diagnosis of schizophrenia according to ICD-10 and DSM-IV criteria.

Exclusion criteria schizophrenic patients:

* Epilepsy or other disorders of the nervous system, further psychiatric or neurological disorders.
* Suicidal tendencies.
* Acute or lifetime alcohol abuse.
* Hearing impairment.
* Intelligence quotient (IQ) below average.
* Non-magnetoencephalography(MEG)/ magnetic resonance imaging(MRI) compatible metallic implants.

Inclusion criteria subjects at risk:

* Signed written informed consent.
* Outpatients of the early diagnosis center of the University Department of Psychiatry at the University Hospital Hamburg-Eppendorf (UKE)Germany.
* Meeting high risk criteria for schizophrenia according to the Structured Interview for Prodromal Syndromes (SIPS).

Exclusion criteria subjects at risk:

* Epilepsy or other disorders of the nervous system, further psychiatric or neurological disorders.
* Suicidal tendencies.
* Acute or lifetime alcohol abuse.
* Hearing impairment.
* IQ below average.
* Non-MEG/MRI compatible metallic implants.

Inclusion criteria healthy controls:

* Signed written informed consent.
* Healthy male and female subjects recruited from students and hospital staff of the University Hospital Hamburg-Eppendorf (UKE), Hamburg, Germany.

Exclusion criteria healthy controls:

* Acute or lifetime psychiatric disorder.
* Suicidal tendencies.
* Epilepsy or other disorders of the nervous system.
* First degree relative with a psychiatric disorder.
* Intake of medication affecting the central nervous system.
* Acute or lifetime alcohol abuse.
* Hearing impairment.
* IQ below average.
* Non-MEG/MRI compatible metallic implants.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Three groups of subjects will be included: patients with a first episode of schizophrenia, subjects at increased risk for schizophrenia, and healthy control subjects.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Brain function | baseline and one-year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Mulert, Prof. Dr., Principal Investigator — University Medical Center Hamburg-Eppendorf, Department of Psychiatry
Locations (1):
- Department of Psychiatry and Psychotherapy, University Hospital Hamburg-Eppendorf (UKE), Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Undecided